CLINICAL TRIAL: NCT02284074
Title: Nasal Lipopolysaccharide (LPS) Challenge in Healthy Volunteers (HVs): Investigation of Tolerability, Dose Response and the Expression Profile of Intercellular Adhesion Molecule-1 (ICAM-1)
Brief Title: Nasal LPS Challenge in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ICRRU/2010/001; 10/H0803/110, ICRRU/2010/001 (Other Grant/Funding Number: CRO1595)
Record Dates: First submitted 2014-09-19; First posted 2014-11-05 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Lipopolysaccharide (LPS); Biomarkers; Chemokines; Cytokines; Gene Expression; Nasal Challenge; Inflammation; Nasal; Nasosorption; Respiratory
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Nasal LPS spray - placebo (Experimental): This is a 5-way crossover, randomised, placebo-controlled study.
  Arms consists of the following nasal challenges:
  placebo, 1, 10, 30 and 100µg LPS.
  Interventions: Other: Nasal LPS spray
- Nasal LPS spray 1µg (Experimental): This is a 5-way crossover, randomised, placebo-controlled study.
  Arms consists of the following nasal challenges:
  placebo, 1, 10, 30 and 100µg LPS.
  Interventions: Other: Experimental: Nasal LPS spray 1µg
- Nasal LPS spray 10 µg (Experimental): This is a 5-way crossover, randomised, placebo-controlled study.
  Arms consists of the following nasal challenges:
  placebo, 1, 10, 30 and 100µg LPS.
  Interventions: Other: Experimental: Nasal LPS spray 10 µg
- Nasal LPS spray 30 µg (Experimental): This is a 5-way crossover, randomised, placebo-controlled study.
  Arms consists of the following nasal challenges:
  placebo, 1, 10, 30 and 100µg LPS.
  Interventions: Other: Experimental: Nasal LPS spray 30 µg
- Nasal LPS spray 100 µg (Experimental): This is a 5-way crossover, randomised, placebo-controlled study.
  Arms consists of the following nasal challenges:
  placebo, 1, 10, 30 and 100µg LPS.
  Interventions: Other: Experimental: Nasal LPS spray 100 µg

INTERVENTIONS:
Other: Nasal LPS spray — LPS solution (250µl) will be prepared at 10, 100, 300 and 1000µg/ml, 100µl is administered to each nostril, both nostrils will be sprayed. The dose per nostril corresponds to 1, 10, 30 and 100µg.
  Arms: Nasal LPS spray - placebo
Other: Experimental: Nasal LPS spray 1µg — LPS solution (250µl) will be prepared at 10, 100, 300 and 1000µg/ml, 100µl is administered to each nostril, both nostrils will be sprayed.
  Arms: Nasal LPS spray 1µg
Other: Experimental: Nasal LPS spray 10 µg — LPS solution (250µl) will be prepared at 10, 100, 300 and 1000µg/ml, 100µl is administered to each nostril, both nostrils will be sprayed.
  Arms: Nasal LPS spray 10 µg
Other: Experimental: Nasal LPS spray 30 µg — LPS solution (250µl) will be prepared at 10, 100, 300 and 1000µg/ml, 100µl is administered to each nostril, both nostrils will be sprayed.
  Arms: Nasal LPS spray 30 µg
Other: Experimental: Nasal LPS spray 100 µg — LPS solution (250µl) will be prepared at 10, 100, 300 and 1000µg/ml, 100µl is administered to each nostril, both nostrils will be sprayed.
  Arms: Nasal LPS spray 100 µg

SUMMARY:
The purpose of this study is to develop a nasal challenge model that causes a mild degree of inflammation, without causing any pain or symptoms, but that allows us to measure a variety of proteins in nasal secretions which causes inflammation in the nose. The nasal challenge model involves spraying the nostrils in the form of a fine mist with 4 different doses (1, 10, 30 and 100µg per nostril) of lipopolysaccharide (LPS) including a placebo. LPS is a type of protein which has been carefully purified from the outer cell wall of certain bacteria, is sterile and does not contain live bacteria, and will not cause infection.

The investigators will measure any inflammation in the nose by looking at cells collected by washing the inside of the nose (nasal lavage) and placing small strips of paper in the nasal cavity. The paper absorbs the nasal fluid and the chemicals produced during inflammation and can be extracted from the paper and analysed in the laboratory. The investigators will also be collecting a small amount of nasal epithelium taken by way of a nasal scrape; this is done by using a Rhinoprobe, a small plastic curette which is used to scrape a small piece of lining of the nose. The investigators hope that information obtained from this study will be used in future studies that will test new study drugs designed to treat diseases of the airways and lungs ( like asthma and chronic obstructive pulmonary disease (COPD) and hay fever.

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODOLOGY This is a single-centre study which will be carried out at the Imperial Clinical Respiratory Research Unit (ICRRU) at St Mary's Hospital in London Paddington.

RECRUITMENT The study will recruit a total of 15 healthy participants.

STUDY VISITS The study will involve a total of 11 outpatients visits. The screening visit is the initial visit where the study is discussed with the participant and written informed consent is obtained by the PI or his designee. This is done prior to performing any study related procedures. The participant will have had the study information sheet for at least 24 hours prior to the visit.

The visit will include the collection of demographic data, height and weight, physical examination by a doctor, medical history, vital signs, body temperature, 12 lead ECG, laboratory assessments (safety bloods) urine drugs of abuse test and pregnancy tests for females. The participant will also be asked to indicate the presence of any nasal symptoms by completing a modified total nasal symptoms score sheet and perform a peak nasal inspiratory flow (PNIF) test.

If eligible, participants will be asked to return for further study visits. Participants will be given 4 different doses of LPS and a placebo in a randomised manner.

There are a total of 5 treatment periods. Each treatment period consists of a 11h visit the first day and a 20 minute visit the following day. There is a total of 12-28 days interval between each treatment period visit.

During the treatment period visits, the study participants will undergo the following study procedures:

1. Nasal lavage to both nostrils and discard with 5ml of 0.9% saline in order to clean the nose prior to nasal LPS challenge.
2. Nasal challenge with LPS (placebo, 1,10, 30 or 100µg per nostril)
3. Nasosorption (right nostril) at -30m, +30m, +1h, then hourly to 10h and 24h
4. Nasal lavage (left nostril) at -30m, +2h, +4h, +8h, +24h
5. Nasal scrape (left nostril) at -30m, +3h, +6h, +24h
6. Modified total nasal symptom score (TNSS) at -30m, +30m, +1h, then hourly to 10h and 24h
7. Peak nasal inspiratory flow (PNIF) rate at -30m, +2h, +4h, +8h, 24h
8. Systemic adverse events
9. Temperature (oral) at -30m, +2h, +4h, +8h
10. Blood pressure and heart rate at -30m
11. Females of child bearing potential will have a pregnancy test performed.

NASAL PROCEDURES IN THE STUDY

1. Nasal washing (nasal lavage): Nasal washings in the nose are carried out by passing a small volume of salt water (saline) fluid into the nose. A nasal adapter shaped like an olive is placed inside the nostril. The participant is then asked to sit forward and the salty water solution (saline) is used to flush in and out of the nose over a one minute period. This procedure is carried out on both nostrils to clean up the nose on the initial study visit and then repeated only on the left nostril on each treatment visit.
2. Nasal lining fluid absorption (nasosorption or SAM): A small strip of absorbent material, that looks and feels like soft tissue paper, will be used to absorb moisture from the inside surface of the nostril. The special absorptive paper will be placed inside the nostril and left for a period of 2 minutes to absorb the nasal lining fluid before being removed, gently sucking up fluid like blotting paper. Putting the paper into the nose can tickle, and cause your eyes to water a little. However, the nasosorption does not hurt and the investigators method has proved to be well tolerated in babies, children and adults. The paper absorbs the nasal fluid and many substances produced by the nasal cells can then be extracted from the paper and measured in the laboratory.
3. Nasal scrape (nasal curettage or Rhinoprobe): A small sterile disposable plastic probe will be inserted into the nose and will be gently pressed against the inside surface lining of the nostril. The 3 inch long probe has a tiny scoop on the end, which can barely be see. 24 tiny samples from each nostril (a pinhead, 2mm, of tissue) will be taken from a part of the nose that has a reduced nerve supply to limit any discomfort. Taking this sample does not cause bleeding, but may cause some mild discomfort, and may make the eyes water slightly. The probe will collect nasal cells from the surface of the nostril which will then be sent for analysis. This method has been performed on many adults, children, and babies, and has been very well tolerated.

STATISTICAL ANALYSIS Each of the measures will be summarised descriptively by dose and time using appropriate summary statistics. If appropriate, response variables will be transformed (e.g. log-transformed). Gene expression data will be normalised by house-keeper gene. The TNSS will be calculated by summing the scores of nasal blockage, nasal discharge/rhinorrhoea, nasal burning/itching/pain sensation, and sneezing at each timepoint. Weighted means of symptom scores will be calculated over the time interval 0 to 10h.

TNSS, nasal sniff pressures, nasosorption measures and gene expression data from the nasal scrapes will each be plotted against time, with a separate plot for each subject and measure, and with LPS dose and placebo represented by separate lines on the plots. Summary statistics (e.g. mean +/- 95% confidence intervals or median and interquartile range) for nasal lavage and gene expression data will be plotted by dose against time.

Correlations will be explored using scatter plots for the following measures:

* Weighted means TNSS vs. maximum TNF-α
* Weighted means TNSS vs. maximum IL-8
* Weighted means TNSS vs. maximum s-ICAM-1
* Maximum ICAM-1 expression vs. maximum TNF-α

Reproducibility of the nasal LPS challenge for ICAM-1 expression and TNF-α will be explored using the following subsets of data:

* Predose data for each period to explore intra-subject variability. Parameter vs. period number will be plotted with a separate line for each subject to explore whether there is a period effect. Box and whisker plots will also be used to summarise the parameter by period.
* Placebo period data - Parameter vs time will be plotted with a separate line for each subject to explore whether there is a time-course effect. Box and whisker plots will also be used to summarise the parameter over time.

Box and whisker plots for ICAM-1 expression and TNF-α and dose and time will be presented to investigate whether these measures return to baseline after 24h.

Additional exploratory analyses may be performed to further characterize the expression profile of ICAM following nasal LPS challenge.

ELIGIBILITY:
INCLUSION CRITERIA

* Males and females aged 18 to 60 years
* Current non-smokers for last 6 months (<5 cigs per week), with a smoking history of <5 pack years
* BMI 20-30 kg/m2

EXCLUSION CRITERIA

* History of allergy
* Upper airway infection in 2 weeks before screening
* Lower respiratory tract infection in past 3 months
* Treatment with local or systemic corticosteroids during previous 2 months
* Signs or symptoms of chronic rhinitis, hypertrophy of turbinates, major septum deviation, nasal polyposis or recurrent sinusitis
* Previous nasal or sinus surgery
* Clinically significant cardiovascular, hepatic, GIT, renal, endocrine, infective, haematological, neurological, dermatological, neoplastic conditions, gastro-oesophageal reflux, depression, TB
* Participation in a therapeutic drug trial in the prior 30 days.
* Medical therapy other than that permitted for contraception.
* Positive pregnancy test
* Inability or unwillingness to use contraception if the patient is a female of child-bearing age.
* History of drug abuse or urine test showing evidence of recreational drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Level of nasal mucosal inter-cellular adhesion molecule-1 (ICAM-1) by gene expression analysis | 8 hours following nasal lipopolysaccharide (LPS) challenge
  Measurement of gene expression (mRNA) for inter-cellular adhesion molecule-1 (ICAM-1) in nasal mucosal curettage samples, 8h following nasal lipopolysaccharide (LPS) challenge.

SECONDARY OUTCOMES:
Nasal mucosal lining fluid IL-1beta levels after nasal lipopolysaccharide (LPS) challenge | Up to 8h after nasal LPS challenge
  Nasal mucosal IL-1beta levels after LPS challenge (area under curve, 0 to 8h) will be compared to placebo responses (AUC, 0-8h) in nasal mucosal lining fluid
Nasal mucosal lining fluid IL-6 levels after nasal lipopolysaccharide (LPS) challenge | Up to 8h after nasal LPS challenge
  Nasal mucosal IL-6 levels after LPS challenge (area under curve, 0 to 8h) will be compared to placebo responses (AUC, 0-8h) in nasal mucosal lining fluid
Nasal mucosal lining fluid CXCL8 levels after nasal lipopolysaccharide (LPS) | Up to 8h after nasal LPS challenge
  Nasal mucosal CXCL8 levels after LPS challenge (area under curve, 0 to 8h) will be compared to placebo responses (AUC, 0-8h) in nasal mucosal lining fluid

CONTACTS AND LOCATIONS:
Overall Officials: Trevor T Hansel, FRCPath, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Respiratory Research Unit (ICRRU), St Mary's Hospital, Paddington, London, United Kingdom

REFERENCES:
- [Background] Barnes PJ. Immunology of asthma and chronic obstructive pulmonary disease. Nat Rev Immunol. 2008 Mar;8(3):183-92. doi: 10.1038/nri2254. Epub 2008 Feb 15. PMID 18274560
- [Background] Anderson GP. Endotyping asthma: new insights into key pathogenic mechanisms in a complex, heterogeneous disease. Lancet. 2008 Sep 20;372(9643):1107-19. doi: 10.1016/S0140-6736(08)61452-X. PMID 18805339
- [Background] Calverley PM, Rennard SI. What have we learned from large drug treatment trials in COPD? Lancet. 2007 Sep 1;370(9589):774-85. doi: 10.1016/S0140-6736(07)61381-6. PMID 17765527
- [Background] Fukata M, Vamadevan AS, Abreu MT. Toll-like receptors (TLRs) and Nod-like receptors (NLRs) in inflammatory disorders. Semin Immunol. 2009 Aug;21(4):242-53. doi: 10.1016/j.smim.2009.06.005. PMID 19748439
- [Background] O'Neill LA, Bryant CE, Doyle SL. Therapeutic targeting of Toll-like receptors for infectious and inflammatory diseases and cancer. Pharmacol Rev. 2009 Jun;61(2):177-97. doi: 10.1124/pr.109.001073. Epub 2009 May 27. PMID 19474110
- [Background] Chanez P, Vignola AM, Vic P, Guddo F, Bonsignore G, Godard P, Bousquet J. Comparison between nasal and bronchial inflammation in asthmatic and control subjects. Am J Respir Crit Care Med. 1999 Feb;159(2):588-95. doi: 10.1164/ajrccm.159.2.9801022. PMID 9927377
- [Background] American Thoracic Society Workshop. Immunobiology of asthma and rhinitis. Pathogenic factors and therapeutic options. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1778-87. doi: 10.1164/ajrccm.160.5.ats7-99. No abstract available. PMID 10556156
- [Background] Linden M, Svensson C, Andersson E, Andersson M, Greiff L, Persson CG. Immediate effect of topical budesonide on allergen challenge-induced nasal mucosal fluid levels of granulocyte-macrophage colony-stimulating factor and interleukin-5. Am J Respir Crit Care Med. 2000 Nov;162(5):1705-8. doi: 10.1164/ajrccm.162.5.9910094. PMID 11069800
- [Background] Alam R, Sim TC, Hilsmeier K, Grant JA. Development of a new technique for recovery of cytokines from inflammatory sites in situ. J Immunol Methods. 1992 Oct 19;155(1):25-9. doi: 10.1016/0022-1759(92)90267-w. PMID 1401965
- [Background] Greiff L, Pipkorn U, Alkner U, Persson CG. The 'nasal pool' device applies controlled concentrations of solutes on human nasal airway mucosa and samples its surface exudations/secretions. Clin Exp Allergy. 1990 May;20(3):253-9. doi: 10.1111/j.1365-2222.1990.tb02680.x. PMID 2364306
- [Background] Howarth PH, Persson CG, Meltzer EO, Jacobson MR, Durham SR, Silkoff PE. Objective monitoring of nasal airway inflammation in rhinitis. J Allergy Clin Immunol. 2005 Mar;115(3 Suppl 1):S414-41. doi: 10.1016/j.jaci.2004.12.1134. PMID 15746881
- [Background] Chawes BL, Edwards MJ, Shamji B, Walker C, Nicholson GC, Tan AJ, Folsgaard NV, Bonnelykke K, Bisgaard H, Hansel TT. A novel method for assessing unchallenged levels of mediators in nasal epithelial lining fluid. J Allergy Clin Immunol. 2010 Jun;125(6):1387-1389.e3. doi: 10.1016/j.jaci.2010.01.039. Epub 2010 Mar 20. No abstract available. PMID 20304470
- [Background] Lin RY, Nahal A, Lee M, Menikoff H. Cytologic distinctions between clinical groups using curette-probe compared to cytology brush. Ann Allergy Asthma Immunol. 2001 Feb;86(2):226-31. doi: 10.1016/S1081-1206(10)62696-8. PMID 11258695
- [Background] Dreskin SC, Dale SN, Foster SM, Martin D, Buchmeier A, Nelson HS. Measurement of changes in mRNA for IL-5 in noninvasive scrapings of nasal epithelium taken from patients undergoing nasal allergen challenge. J Immunol Methods. 2002 Oct 15;268(2):189-95. doi: 10.1016/s0022-1759(02)00206-5. PMID 12215387
- [Background] Proud D, Turner RB, Winther B, Wiehler S, Tiesman JP, Reichling TD, Juhlin KD, Fulmer AW, Ho BY, Walanski AA, Poore CL, Mizoguchi H, Jump L, Moore ML, Zukowski CK, Clymer JW. Gene expression profiles during in vivo human rhinovirus infection: insights into the host response. Am J Respir Crit Care Med. 2008 Nov 1;178(9):962-8. doi: 10.1164/rccm.200805-670OC. Epub 2008 Jul 24. PMID 18658112
- [Background] Jalowayski AA, Walpita P, Puryear BA, Connor JD. Rapid detection of respiratory syncytial virus in nasopharyngeal specimens obtained with the rhinoprobe scraper. J Clin Microbiol. 1990 Apr;28(4):738-41. doi: 10.1128/jcm.28.4.738-741.1990. PMID 2185261
- [Background] Erin EM, Neighbour H, Tan AJ, Min Kon O, Durham SR, Hansel TT. Nasal testing for novel anti-inflammatory agents. Clin Exp Allergy. 2005 Aug;35(8):981-5. doi: 10.1111/j.1365-2222.2005.02311.x. No abstract available. PMID 16120078
- [Background] Singh J, Schwartz DA. Endotoxin and the lung: Insight into the host-environment interaction. J Allergy Clin Immunol. 2005 Feb;115(2):330-3. doi: 10.1016/j.jaci.2004.11.021. PMID 15696090
- [Background] Peden DB, Tucker K, Murphy P, Newlin-Clapp L, Boehlecke B, Hazucha M, Bromberg P, Reed W. Eosinophil influx to the nasal airway after local, low-level LPS challenge in humans. J Allergy Clin Immunol. 1999 Aug;104(2 Pt 1):388-94. doi: 10.1016/s0091-6749(99)70383-0. PMID 10452761
- [Background] Bals R. Lipopolysaccharide and the lung: a story of love and hate. Eur Respir J. 2005 May;25(5):776-7. doi: 10.1183/09031936.05.00025405. No abstract available. PMID 15863630
- [Background] Danuser B, Rebsamen H, Weber C, Krueger H. Lipopolysaccharide-induced nasal cytokine response: a dose-response evaluation. Eur Arch Otorhinolaryngol. 2000 Dec;257(10):527-32. doi: 10.1007/s004050000285. PMID 11195030
- [Background] Sigsgaard T, Bonefeld-Jorgensen EC, Kjaergaard SK, Mamas S, Pedersen OF. Cytokine release from the nasal mucosa and whole blood after experimental exposures to organic dusts. Eur Respir J. 2000 Jul;16(1):140-5. doi: 10.1034/j.1399-3003.2000.16a25.x. PMID 10933100
- [Background] Nita I, Hollander C, Westin U, Janciauskiene SM. Prolastin, a pharmaceutical preparation of purified human alpha1-antitrypsin, blocks endotoxin-mediated cytokine release. Respir Res. 2005 Jan 31;6(1):12. doi: 10.1186/1465-9921-6-12. PMID 15683545
- [Background] Bachar O, Gustafsson J, Jansson L, Adner M, Cardell LO. Lipopolysaccharide administration to the allergic nose contributes to lower airway inflammation. Clin Exp Allergy. 2007 Dec;37(12):1773-80. doi: 10.1111/j.1365-2222.2007.02842.x. Epub 2007 Oct 17. PMID 17941911
- [Background] Ekman AK, Fransson M, Rydberg C, Adner M, Cardell LO. Nasal challenge with LPS stimulates the release of macrophage inflammatory protein 1alpha. Int Arch Allergy Immunol. 2009;149(2):154-60. doi: 10.1159/000189199. Epub 2009 Jan 6. PMID 19127073
- [Background] Mayr FB, Spiel A, Leitner J, Marsik C, Germann P, Ullrich R, Wagner O, Jilma B. Effects of carbon monoxide inhalation during experimental endotoxemia in humans. Am J Respir Crit Care Med. 2005 Feb 15;171(4):354-60. doi: 10.1164/rccm.200404-446OC. Epub 2004 Nov 19. PMID 15557136
- [Background] Michel O, Dentener M, Cataldo D, Cantinieaux B, Vertongen F, Delvaux C, Murdoch RD. Evaluation of oral corticosteroids and phosphodiesterase-4 inhibitor on the acute inflammation induced by inhaled lipopolysaccharide in human. Pulm Pharmacol Ther. 2007;20(6):676-83. doi: 10.1016/j.pupt.2006.08.002. Epub 2006 Sep 14. PMID 17045826
- [Background] Fijen JW, Kobold AC, de Boer P, Jones CR, van der Werf TS, Tervaert JW, Zijlstra JG, Tulleken JE. Leukocyte activation and cytokine production during experimental human endotoxemia. Eur J Intern Med. 2000 Apr;11(2):89-95. doi: 10.1016/s0953-6205(00)00068-6. PMID 10745152
- [Background] Michel O, Murdoch R, Bernard A. Inhaled LPS induces blood release of Clara cell specific protein (CC16) in human beings. J Allergy Clin Immunol. 2005 Jun;115(6):1143-7. doi: 10.1016/j.jaci.2005.01.067. PMID 15940126
- [Background] Michel O, Nagy AM, Schroeven M, Duchateau J, Neve J, Fondu P, Sergysels R. Dose-response relationship to inhaled endotoxin in normal subjects. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 1):1157-64. doi: 10.1164/ajrccm.156.4.97-02002. PMID 9351616
- [Background] Nightingale JA, Rogers DF, Hart LA, Kharitonov SA, Chung KF, Barnes PJ. Effect of inhaled endotoxin on induced sputum in normal, atopic, and atopic asthmatic subjects. Thorax. 1998 Jul;53(7):563-71. doi: 10.1136/thx.53.7.563. PMID 9797755
- [Derived] Dhariwal J, Kitson J, Jones RE, Nicholson G, Tunstall T, Walton RP, Francombe G, Gilbert J, Tan AJ, Murdoch R, Kon OM, Openshaw PJ, Hansel TT. Nasal Lipopolysaccharide Challenge and Cytokine Measurement Reflects Innate Mucosal Immune Responsiveness. PLoS One. 2015 Sep 14;10(9):e0135363. doi: 10.1371/journal.pone.0135363. eCollection 2015. PMID 26367003